CLINICAL TRIAL: NCT07267208
Title: A Prospective Study to Evaluate the Efficacy and Safety of Entecavir ODT Conversion in Stable Liver Transplant Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jongman Kim (Other)
Responsible Party: Sponsor-Investigator, Jongman Kim, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025-09-055
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hepatitis B Virus; Liver Transplant
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Entecavell ODT (Experimental): Entecavir ODT is administered once every day with 0.5mg PO
  Interventions: Drug: Entecavell ODT

INTERVENTIONS:
Drug: Entecavell ODT — Entecavir ODT is administered once every day with 0.5mg PO for 48 weeks.

SUMMARY:
This clinical study aims to evaluate the efficacy and safety of switching to entecavir orally disintegrating tablets (ETV-ODT) in liver transplant recipients with chronic hepatitis B, with a particular focus on the impact of the conversion on renal function.

After providing written informed consent, participants will undergo screening assessments to determine eligibility based on the inclusion and exclusion criteria. Eligible participants who receive the investigational product will visit the study site at predetermined time points over a 48-week period to complete the scheduled study procedures.

DETAILED DESCRIPTION:
This study aims to evaluate the antiviral efficacy, safety, and potential improvement in medication adherence after converting stable liver transplant recipients to Entecabell ODT. Only participants who meet all inclusion and exclusion criteria will receive the investigational product. After conversion, participants will take Entecabell ODT 0.5 mg once daily for 48 weeks and will be followed according to the scheduled visits and assessments.

The primary objective of the study is to assess the impact of switching from entecavir tablets to Entecabell ODT on renal function in liver transplant recipients receiving entecavir for HBV prophylaxis. Secondary objectives include evaluating the antiviral effect against HBV and the potential improvement in medication adherence following conversion to Entecabell ODT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 years or older.
2. Patients who have maintained stable liver graft function for one year after liver transplantation due to HBV and meet the following conditions:

   1. AST and ALT < 35IU/L
   2. HBsAg: Negative
   3. HBV DNA: Not detected
3. Patients who have been taking entecavir for HBV prophylaxis for at least 1 year.
4. Patients with a tacrolimus trough level maintained between 3-10 ng/mL. 5 .Patients who have voluntarily decided to participate in the clinical trial after fully understanding the detailed explanation of the trial and have provided written consent.

Exclusion Criteria:

1. Patients who have undergone transplantation of organs other than the liver or re-transplantation.
2. Patients who have received bioartificial liver system treatment or auxiliary partial orthotopic liver transplantation (APOLT) before the transplantation.
3. Patients with concurrent viral infections (HCV, HIV).
4. Patients with eGFR <30 or those undergoing dialysis
5. Pregnant or breastfeeding women.
6. Patients or their spouses/partners who do not agree to use medically acceptable and appropriate contraception methods* during the clinical trial period.

   * Appropriate contraception methods: hormonal contraception, intrauterine device (IUC or IUS), tubal ligation, tubal occlusion, hysterectomy, vasectomy, double barrier methods (combined use of male or female condoms with cervical caps, diaphragms, or contraceptive sponges), single barrier methods with spermicide.
7. Patients with a history of hypersensitivity to Entecavir.
8. Patients who are deemed unsuitable for participation in the clinical trial by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in eGFR at week 48 | Baseline to week 48
  Change in eGFR from baseline to week 48 following ETV-ODT conversion

SECONDARY OUTCOMES:
Change in Creatinine, cystatin C profile | Baseline to week 48
  Change in Creatinine, cystatin C profile from baseline to week 48 following ETV-ODT conversion
Change in CKD stage | Baseline to week 48
  Change in the proportion of participants by CKD stage from baseline to Week 48 following ETV-ODT conversion
Incidence of HBV recurrence | Baseline to week 48
  Incidence of HBV recurrence
Change in cholesterol status, proteinuria and liver stiffness | Baseline to week 48
  Change in cholesterol status (LDL, HDL, total cholesterol, triglycerides), proteinuria (protein-to-creatinine ratio and albumin-to-creatinine ratio), and liver stiffness by FibroScan from baseline to Week 48 following ETV-ODT conversion
Change in medication adherence | Baseline to week 48
  Change in medication adherence from baseline to Week 48 following ETV-ODT conversion
Incidence of graft failure and mortality | Baseline to week 48
  Incidence of graft failure and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jongman Kim, Ph, MD, Principal Investigator — Samsung Medical Center